CLINICAL TRIAL: NCT00517049
Title: A Phase II, Single-Arm, Open-Label Study of the Safety, Pharmacokinetics, and Efficacy of Multiple Doses of PRO95780 Administered Intravenously in Combination With Rituximab in Patients With Follicular, CD20-Positive B-Cell Non-Hodgkin's Lymphoma That Has Progressed Following Previous Rituximab Therapy
Brief Title: A Study of PRO95780 in Combination With Rituximab in Patients With Non-Hodgkin's Lymphoma That Has Progressed Following Previous Rituximab Therapy (APM4083g)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APM4083g
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: NHL; Rituxan; Lymphoma; CD20-positive; B-Cell; APM4083g
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — drozitumab; Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PRO95780; Drug: rituximab

INTERVENTIONS:
Drug: PRO95780 — Intravenous repeating dose
Drug: rituximab — Intravenous repeating dose

SUMMARY:
This Phase II, single-arm, open-label, multicenter trial is designed to evaluate the safety, efficacy, and pharmacokinetics of PRO95780 when combined with rituximab in patients with follicular, CD20-positive B-cell NHL that has progressed following previous rituximab therapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥ 18 years
* Diagnosis of follicular, CD20-positive B-cell NHL
* Progression of disease after an objective response or stable disease lasting > 6 months following completion of the most recent rituximab-containing regimen
* Measurable disease
* Life expectancy of > 3 months

Exclusion Criteria:

* Grade 3b follicular lymphoma (according to the WHO classification) or histologic transformation from follicular lymphoma to aggressive lymphoma
* Prior radiotherapy to a lesion(s) that will be used to assess response unless that lesion(s) shows clear evidence of lymphoma progression at baseline
* Radiotherapy to a peripheral lesion within 14 days prior to Cycle 1, Day 1 or radiotherapy to a thoracic, abdominal, or pelvic field within 28 days prior to Cycle 1, Day 1
* Concurrent systemic corticosteroid therapy
* Other invasive malignancies within 3 years prior to first study drug administration except for adequately treated basal or squamous cell skin cancer, in situ carcinoma of the cervix, in situ breast cancer, in situ prostate cancer, limited-stage bladder cancer, or other cancers from which the patient has been disease-free for at least 3 years.
* History or evidence on physical examination of central nervous system (CNS) disease
* Prior treatment with agonistic DR4 or DR5 antibodies or Apo2L/TRAIL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-03 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Objective response, as determined by independent review facility | 8 months

SECONDARY OUTCOMES:
Progression-free survival, as determined by independent review facility | up to 12 months
Duration of objective response, as determined by independent review facility | up to 10.3 months
Overall survival | Up to 18.5 months
Objective response, as determined by the investigator | Up to 8 months
Progression-free survival, as determined by the investigator | Up to 18.5 months
Duration of objective response, as determined by the investigator | Up to 14.1 months

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Bray, M.D., Study Director — Genentech, Inc.